CLINICAL TRIAL: NCT03921892
Title: A Randomized Feasibility and Acceptability Study Comparing In-person to On-line Parenting Education for Adolescent Fathers
Brief Title: A Comparison of Parenting Education Approaches for Adolescent Fathers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Rita Sue Lasiter, Principal Investigator, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019000019
Record Dates: First submitted 2019-04-14; First posted 2019-04-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Adolescent, Parenting

STUDY DESIGN:
Intervention Model Description: Using a block randomization generator, participants will be randomized into either in-person or on-line parenting education that will take place over a two week period of time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person parenting education (Other): Participants will complete two six-hour in-person parenting education sessions on two consecutive Saturdays
  Interventions: Behavioral: Parenting Education
- On-line parenting education (Active Comparator): Participants will complete on-line parenting education at the times and locations of their choice over a two-week period.
  Interventions: Behavioral: Parenting Education

INTERVENTIONS:
Behavioral: Parenting Education — Parenting education such as positive parenting interactions with their child, knowledge of developmental milestones and interactions with the child to support that development, as well as co-parenting skills will be provided either in-person or on-line to adolescent fathers

SUMMARY:
This feasibility and acceptability study will compare in-person to web-based parenting education for adolescent fathers on the outcomes of parenting confidence and participation in parenting activities.

DETAILED DESCRIPTION:
This is a randomized feasibility and acceptability study using a block generator for randomization of participants aged 15 to 21 into either in-person parenting education or on-line parenting. Outcome measures include parenting self-efficacy and participation in daily parenting activities. Participants will take part in approximately twelve hours of parenting education, whether in-person or on-line. Recruitment flyers will be placed in two primary care clinics and a large regional hospital's Labor & Delivery and Postpartum (Mother-Baby) Units. Participants will seek out the opportunity to participate by calling the phone number or sending an e-mail to the investigators to learn more about the study and their potential participation. If participants meet eligibility criteria and elect to participate, baseline measurements will be completed after enrollment, with follow-up measures at one month and two months.

ELIGIBILITY:
Inclusion Criteria:

* age 15 to 21,
* be able to read and understand English (as determined by having the individual read a brief, eighth grade reading level paragraph),
* able to begin the intervention within six weeks of their infant's birth,
* be able to participate in an intervention over two weeks, requiring approximately a 12-hour time commitment: either in-person on two Saturdays for six hours each, or a self-paced content of videos and resource materials over two weeks,
* own or have access to a device with internet access and
* have a working e-mail address.

Exclusion Criteria:

* Any condition that might prevent the father's infant from reaching normal developmental milestones will participation, including congenital malformations or prematurity requiring prolonged/ ongoing infant hospitalization.

Ages: 15 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Adolescent males aged 15 to 21
Enrollment: 10 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Feasibility Measure 1 | 12 months
  Did recruitment numbers meet goals
Feasibility Measure 2 | 12 months
  Attrition rate of participants
Feasibility Measure 3 | 12 months
  Percent of data missing from data collection tools
Acceptability Survey Measure 1 (Likert Scale) | 12 months
  Acceptability of learning content to participants
Acceptability Survey Measure 2 (Likert Scale) | 12 months
  Acceptability of time burden to participants
Acceptability Survey Measure 3 (Likert Scale) | 12 months
  Acceptability of learning method to participants

SECONDARY OUTCOMES:
What is the difference between in-person education as compared to on-line parenting education on parental self-efficacy of adolescent fathers as measured by the Parenting Sense of Competence Scale (PSOC)? | 12 months
  Does providing parenting education to adolescent fathers, either in-person or on-line, change their levels of parenting self-efficacy
What is the difference between in-person parenting education as compared to on-line parenting education on participation in parenting activities of adolescent fathers as measured by the Child Care Activities Scale (CCAS)? | 12 months
  Does either in-person or on-line parenting education impact the participation in parenting activities of adolescent fathers?

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Anchorage Neighborhood Health Center, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Family Medicine Clinic, Anchorage, Alaska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savio Beers LA, Hollo RE. Approaching the adolescent-headed family: a review of teen parenting. Curr Probl Pediatr Adolesc Health Care. 2009 Oct;39(9):216-33. doi: 10.1016/j.cppeds.2009.09.001. PMID 19857857
- [Background] Kiselica, M. S., & Kiselica, A. M. (2014). The complicated worlds of adolescent fathers: Implications for clinical practice, public policy, and research. Psychology of Men & Masculinity, 15(3), 260-274. doi:10.1037/a0037043
- [Background] Sevigny PR, Loutzenhiser L. Predictors of parenting self-efficacy in mothers and fathers of toddlers. Child Care Health Dev. 2010 Mar;36(2):179-89. doi: 10.1111/j.1365-2214.2009.00980.x. Epub 2009 Jul 23. PMID 19645829
- [Background] Seymour, M., Dunning, M., Cooklin, A., & Giallo, R. (2014). Socioecological factors associated with fathers' well-being difficulties in the early parenting period. Clinical Psychologist, 18(2), 63-73. doi:10.1111/cp.12016
- [Background] Wilkes L, Mannix J, Jackson D. 'I am going to be a dad': experiences and expectations of adolescent and young adult expectant fathers. J Clin Nurs. 2012 Jan;21(1-2):180-8. doi: 10.1111/j.1365-2702.2011.03715.x. Epub 2011 Jun 5. PMID 21645156
- [Background] Rominov H, Giallo R, Whelan TA. Fathers' postnatal distress, parenting self-efficacy, later parenting behavior, and children's emotional-behavioral functioning: A longitudinal study. J Fam Psychol. 2016 Dec;30(8):907-917. doi: 10.1037/fam0000216. Epub 2016 May 16. PMID 27183189
- [Background] Love SM, Sanders MR, Turner KM, Maurange M, Knott T, Prinz R, Metzler C, Ainsworth AT. Social media and gamification: Engaging vulnerable parents in an online evidence-based parenting program. Child Abuse Negl. 2016 Mar;53:95-107. doi: 10.1016/j.chiabu.2015.10.031. Epub 2016 Feb 12. PMID 26880281
- [Background] Hall CM, Bierman KL. Technology-assisted Interventions for Parents of Young Children: Emerging Practices, Current Research, and Future Directions. Early Child Res Q. 2015 4th Quarter;33:21-32. doi: 10.1016/j.ecresq.2015.05.003. Epub 2015 May 23. PMID 27773964
- [Background] Fagan, J., Bernd, E., & Whiteman, V. (2007). Adolescent fathers' parenting stress, social support, and involvement with infants. Journal of Research on Adolescence, 17(1), 1-22. doi:10.1111/j.1532-7795.2007.00510.x
- [Result] Cronenwett LR, Sampselle CM, Wilson WR. The Child Care Activities Scale and Parental Role Preference Scale. Res Nurs Health. 1988 Oct;11(5):301-8. doi: 10.1002/nur.4770110505. PMID 3175054
- [Result] Johnston, C., & Mash, E. J., (1989). A measure of parenting satisfaction and efficacy. Journal of Clinical Child Psychology, 18(2), 167-175